CLINICAL TRIAL: NCT06461286
Title: A Phase 1a Open-Label, Single Ascending Dose Study to Evaluate the Safety and Tolerability of Intravitreally Administered PYC-001 in Participants With Confirmed OPA1 Mutation-Associated Autosomal Dominant Optic Atrophy
Brief Title: SAD of IVT PYC-001 in OPA1 Mutation-Associated Autosomal Dominant Optic Atrophy (Sundew)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PYC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PYC-001-101
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: OPA1 Gene Mutation; Autosomal Dominant Optic Atrophy; Hereditary Optic Atrophies; Kjer Optic Atrophy
MeSH Terms: conditions — Optic Atrophy, Autosomal Dominant; Optic Atrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm dose escalation study of PYC-001 (Experimental): Drug: PYC-001
  Phase 1a Open-Label, Single Ascending Dose Study to Evaluate the Safety and Tolerability of Intravitreally Administered PYC-001 in participants with Confirmed OPA1 Mutation-Associated Autosomal Dominant Optic Atrophy
  Interventions: Drug: PYC-001

INTERVENTIONS:
Drug: PYC-001 — Single Group Assignment

SUMMARY:
A First-in-Human multi-centre, prospective, Phase1a, Single Ascending Dose (SAD) interventional study of PYC-001 in participants with confirmed OPA1 mutation (haploinsufficiency) associated ADOA.

DETAILED DESCRIPTION:
This is a First-In-Human multi-centre, prospective, Phase 1a, single ascending dose (SAD) interventional study of PYC-001 in participants with confirmed OPA1 mutation (haploinsufficiency) associated ADOA.

Following confirmation of eligibility on Day-1, one(1) eye will be selected for study participation (the "study eye"), and the other eye will be designated as the "fellow eye". Selection of the "Study eye" will be the eye with worse vision. If both eyes have similar visual acuity and visual field information, the choice of study eye will be determined at the discretion of the Investigator in consultation with the participant.

Each eligible participant will receive a single intravitreal (IVT) injection of PYC-001 in their study eye on Day 1, and will be monitored for dose limiting toxicities (DLTs) for 4 weeks. The study will use a 3+3 escalation scheme and will involve up to three PYC-001 dose groups. Cohorts of 3 participants will be initially enrolled at each dose level, and then expanded to 6 participants per cohort in the event of a DLT or any >> Grade 2 adverse events (AEs) that are deemed related to study treatment. Within each cohort, dosing will be staggered with a 7-day interval between the first participant receiving investigational product (IP), PYC-001, and the remaining 2 participants receiving IP.

If >> 2 DLTs are observed in 6 participants in any cohort, and the previous lower dose cohort was not previously expanded to 6 participants per the 3+3 design rules, the lower dose cohort will be expanded to include evaluation of 6 participants. If this lower dose level has << 1 DLTs it will be considered the maximum tolerated dose (MTD). Alternatively, a dose half-way between the previous lower dose, and the dose with >> 2 participants showing DLTs may be selected for evaluation.

If no DLTs or any >> Grade 2 AEs are observed in the first 3 participants treated within a cohort, then escalation to the next dose cohort can proceed following review of the collated 4-week safety data by the safety review committee (SRC).

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects;
2. Adult males and females, aged 18 years and above at screening;
3. Body mass index (BMI) ≥18.0 and ≤32.0 kg/m2, with a body weight ≤ 100kg at screening;
4. Have a molecular (genetic) diagnosis of OPA1 mutation at screening;
5. Have a clinical diagnosis of OPA1 mutation-associated ADOA at screening;
6. Participants with BCVA of between 20/40 (70 ETDRS letters) and 20/160 (39-43 ETDRS letters). If both eyes meet this eligibility criteria, the eye with worse BCVA will be selected as the study eye and the other eye will be designated as the "fellow eye";
7. Medically healthy (in the opinion of the Investigator), as determined by pre-study medical history, and without clinically significant abnormalities including:

   1. Physical examination without any clinically relevant findings;
   2. Systolic BP in the range of 90 to 160mmHg and diastolic BP in the range of 50 to 95 mmHg after 5 minutes in supine of semi-supine position;
   3. Heart rate in the range of 45 to 100 bpm after 5 minutes rest in supine or semi-supine position;
   4. Body temperature (tympanic), between 35.5°C and 37.7°C;
   5. ECG without clinically significant abnormalities including QT interval corrected for Fredericia (QTcF) < 450 msec for male subjects and < 470 msec for female subjects;
   6. No clinically significant findings in clinical chemistry, hematology, coagulation and urinalysis tests at screening.
8. Female volunteers must be of non-child-bearing potential, i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the screening visit) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle stimulating hormone [FSH] level consistent with postmenopausal status, per local laboratory guidelines). Females receiving hormone replacement therapy (HRT) may be considered for inclusion if the need for HRT is for no other medical reason than to treat symptoms associated with menopause. If female participants are of child-bearing potential, they must:

   1. Have a negative pregnancy test at the screening visit, on study Day -1 and study Day 1 prior to dosing;
   2. Agree not to attempt to become pregnant or donate ova from signing the consent form until at least 130 days after IVT administration of PYC-001 and at least 30 days after the final dose of ANX776;
   3. Agree to use adequate contraception (defined as use of a condom by the male partner combined with use of a highly effective method of contraception from one month prior to screening until at least 30 days after the final dose of ANX776 (study Day 336), if not exclusively in a same-sex relationship or abstinent as a committed lifestyle.
9. Male volunteers must:

   1. Agree not to donate sperm from signing the consent form until at least 190 days after IVT administration of PYC-001 and at least 90 days after the final dose of ANX776;
   2. If engaging in sexual intercourse with a female partner who could become pregnant, agree to use adequate contraception (defined as use of a condom combined with use of a highly effective method of contraception) from signing the consent form until at least 190 days after IVT administration of PYC-001 and at least 90 days after the final dose of ANX776;
   3. If engaging in sexual intercourse with a female partner who is not of child-bearing potential or a same-sex partner, agree to use a condom from signing the consent form until at least 190 days after IVT administration of PYC-001 and at least 90 days after the final dose of ANX776;
10. Have suitable venous access for blood sampling
11. Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. Participants has a known allergy to PYC-001 or any of its excipients;
2. Demonstrated clinically significant co-morbidities, which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial and/or confound study outcomes;
3. Females who are breastfeeding or planning to breastfeed;
4. Have mutations in genes that cause ADOA, other than OPA1 (for example in case of dominant negative ADOA) and ADOA Plus;
5. Have received any prior cell or gene therapy for a retinal condition;
6. Within 3 months prior to study Day -1, have undergone any vitreoretinal surgery (scleral buckle, pars plana vitrectomy, retrieval of a dropped nucleus or intraocular lens, radial optic neurotomy, sheathotomy, cyclodestructive procedures or multiple filtration surgeries [2 or more]) or any other ocular surgery;
7. Within 3 months prior to study Day -1, have placement of an Ozurdex® implant;
8. Within 3 months prior to study Day -1 have placement of Retisert® of Iluvien® implants;
9. Have ocular media opacity or poor pupillary dilation prohibiting quality ophthalmic evaluation or photography, as assessed by the Investigator;
10. Macular edema (intraretinal, sub-retinal or other fluid) requiring regular treatment at a frequency of less than every 6 weeks; macular edema must be stable for at least 3 months prior to screening. Note, the above conditions will be permitted for inclusion if, in the opinion of the Investigator and in consultation with the SMM, they will not interfere with study evaluations, or have resolved by study Day -1 prior to dose administration;
11. Have used any investigational drug or device within 90 days or 5 estimated half-lives of the investigational drug or device (whichever is longer) prior to study Day -1, or plan to participate in another study of a drug or device during the study period. Participation in observational trials is allowed based on Investigator discretion and consultation with the Sponsor's Medical Representative;
12. Have a recent history (< 6 months) of or current excessive recreational drug or alcohol use, in the opinion of the Investigator. Note: excessive alcohol use is defined as regular consumption of > 10 standard drinks per week or > 4 standard drinks per day, where 1 standard drink is defined as 10 grams of pure alcohol;
13. Positive alcohol breath test as assessed at screening, and on study Day -1 and study Day 1;
14. Positive urine drugs of abuse as assessed at screening and on study Day -1 and study Day 1;
15. Any retinal pathology other than ADOA or any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence, type, severity and relationship of ocular treatment-emergent adverse events (TEAEs), and treatment-emergent serious adverse events (SAEs) in the study eye | 24 weeks
Incidence, type, severity and relationship of ocular treatment-emergent adverse events (TEAEs), and treatment-emergent serious adverse events (SAEs) in the study eye | 48 weeks
Incidence, type, severity and relationship of ocular TEAEs, and treatment-emergent SAEs in the fellow eye | 24 weeks
Incidence, type, severity and relationship of ocular TEAEs, and treatment-emergent SAEs in the fellow eye | 48 weeks
Incidence, type, severity and relationship of non-ocular TEAEs, and treatment-emergent SAEs | 24 weeks
Incidence, type, severity and relationship of non-ocular TEAEs, and treatment-emergent SAEs | 48 weeks
Change from baseline for vital signs measurements (heart rate [HR], systolic and diastolic blood pressure [BP], tympanic temperature, respiratory rate [RR]) | 48 weeks
Change from baseline for 12-lead electrocardiogram (ECG) parameters | 48 weeks
  Twelve-lead ECG (including but not limited to the measurements of ventricular HR, PR interval, QRS duration, QT interval and QtcF) will be performed. ECGs will be performed in triplicate at screening only with each replicate separated by at least 1 minute and the full set of triplicates completed within 5 minutes. The mean value for the triplicate will be utilized. Single ECGs will be collected at all other timepoints.
Change from baseline for clinical laboratory results - hematology | 48 weeks
  Hematology Screening parameters: Hematocrit, Hemoglobin, Mean Corpuscular hemoglobin, mean corpuscular hemoglobin concentration, mean corpuscular volume, mean platelet volume, packed cell volume, platelet count, red blood cell count, reticulocyte count, white blood cell count with differential neutrophil count, eosinophil count, basophil count, lymphocyte count, monocyte count.
Change from baseline for clinical laboratory results - clinical chemistry | 48 weeks
  Clinical Chemistry screening parameters: Albumin, alkaline phosphatase, alanine aminotransferase, amylase, anion gap, aspartate aminotransferase, bicarbonate, calcium, ionized calcium, chloride, conjugated (direct) and unconjugated bilirubin, creatinine, eGFR, Creatinine kinase, Gamma glutamyl transferase, Globulin, Glucose, High density lipoprotein, Lactate dehydrogenase, Lipase, Low density lipoprotein, Magnesium, Phosphate, Potassium, Sodium, Total bilirubin, Total cholesterol, Total protein, Triglycerides, Urate, Urea
Change from baseline for clinical laboratory results - coagulation | 48 weeks
  Coagulation screening parameters: Activated partial thromboplastin time, International normalized ratio/Prothrombin time, Fibrinogen
Change from baseline for clinical laboratory results - urinalysis | 48 weeks
  Urinalysis screening parameters: Bilirubin, Blood, Glucose, Ketones, Leukocyte esterase, Nitrites, pH, Protein, Specific gravity, Urobilinogen

SECONDARY OUTCOMES:
Change from baseline for Best-corrected visual acuity (BCVA) letter score using Early Treatment of Diabetic Retinopathy Study(ETDRS) | Week 4, Week 12, Week 24, Week 48
Change from baseline for Low contrast visual acuity (LCVA) | Week 4, Week 12, Week 24, Week 48
Change from baseline for Perimetry | Week 4, Week 12, Week 24, Week 48
Change from baseline for posterior eye healthy by fundus examination, using ultrawide funduscopy | Week 4, Week 12, Week 24, Week 48
Change from baseline for color vision by Hardy Rand Rittler test | Week 4, Week 12, Week 24, Week 48
Change from baseline for contrast sensitivity by Pelli Robson Chart | Week 4, Week 12, Week 24, Week 48
Change from baseline for visual field sensitivity by Static Perimetry | Week 4, Week 12, Week 24, Week 48
Change from baseline for Multifocal Visual Evoked Potential (mfVEP) | Week 4, Week 12, Week 24, Week 48
Change from baseline for retinal nerve fiber layer (RNFL) and Ganglion Cell Layer (GCL) thickness by Spectral domain optical coherence tomography (SD-OCT) | Week 4, Week 12, Week 24, Week 48
Change from baseline for mitochondrial function test by flavoprotein fluorescence (FPF) analyzer (Ocumet Beacon) | Week 4, Week 12, Week 24, Week 48
Change from baseline for Detection of Apoptosis in Retinal Cells (DARC) | Week 4, Week 12, Week 24, Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Sreenivasu Mudumba, PhD, Study Chair — PYC Therapeutics
Locations (2):
- Australia (2):
  - Save Sight Institute - Sydney Eye Hospital, Sydney, New South Wales
  - Center for Eye Research Australia (CERA), East Melbourne, Victoria